CLINICAL TRIAL: NCT01826578
Title: Prospective Randomized Controlled Trial to Analyze the Benefits of Single Port Laparoscopic Myomectomy in the View of Cosmetics and Patient Satisfaction
Brief Title: Single Port Myomectomy Versus Conventional Myomectomy
Acronym: SM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, JungRyoel Lee, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jrlee01
Record Dates: First submitted 2013-03-22; First posted 2013-04-08 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Cosmetic Outcomes
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single port arm (Experimental)
  Interventions: Procedure: using only one port for laparoscopic surgery
- Conventional arm (No Intervention): Using 3-4 port for laparosocpic surgery

INTERVENTIONS:
Procedure: using only one port for laparoscopic surgery — using only one port for laparoscopic surgery
  Other Names: Single port intervention
  Arms: single port arm

SUMMARY:
This study is about the evaluation of which benefits single port laparoscopic myomectomy has in the perspective of cosmetics and patient satisfaction.

DETAILED DESCRIPTION:
There were several studies about feasibility and cosmetic benefit of single port laparoscopic adnexal surgery and hysterectomy compared to conventional multiport laparoscopic surgery. Meanwhile, no study mentioned benefit of single port laparoscopic surgery in myomectomy because single port myomectomy needs more labor and operator's skill than other pelvic surgery. At this point, the investigators need to verify the effectiveness and benefit of single port laparoscopic myomectomy.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal women
* image confirmed myoma
* scheduled to have laparoscopic myomectomy
* number of myoma =<4 and largest size <10cm

Exclusion Criteria:

* scheduled to have co-operation of other surgery
* clinically significant hematologic abnormality
* DM or malnutrition
* under the medication which can affect wound healing
* previous history of other pelvic surgery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Cosmetic benefits of single port laparoscopic myomectomy to conventional myomectomy in the view of scar evaluation | for 8 weeks
  The characteristics of scar such as color, pliability, and stiffness are willing to be measured in 1 week and 8 week later after myomectomy. The level of satisfaction of patients will also be evaluated.
Cosmetic benefits of single port laparoscopic myomectomy to conventional myomectomy in the view of patient satisfaction | for 8 weeks
  Patient satisfaction about scar formation after myomectomy are willing to be evaluated after surgery.

SECONDARY OUTCOMES:
General composite characteristics of surgery procedure and outcome | 1 week
  Composite parameters about surgery outcome and complication such as Op time, Drop of Hb, postop pain, duration of hospital stay, intraop complication, postop complication are willing to be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul University Bundang Hospital OB & GY, Sungnam-si, Kyeonggi-do, South Korea